CLINICAL TRIAL: NCT00247650
Title: Randomized Multi-Center Study Comparing Prolonged Primary Systemic Endocrine Therapy With Letrozole Alone or in Combination With Zoledronic Acid in Early Breast Cancer (NEOadjuvant Study in CANada)
Brief Title: Comparison Study of Letrozole Alone or Letrozole With Zoledronic Acid in Early Breast Cancer, Neoadjuvant Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446GCA08
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2009-11

CONDITIONS: Breast Cancer
Keywords: neoadjuvant, postmenopausal women, breast cancer, hormonal therapy, bisphosphonate
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid; Letrozole

INTERVENTIONS:
Drug: Zoledronic Acid; Letrozole

SUMMARY:
This study is to measure the extent of tumor shrinkage when Letrozole and Zoledronic Acid are given before surgery to newly diagnosed post-menopausal women with early breast cancer

ELIGIBILITY:
Inclusion Criteria

* Postmenopausal women
* Newly diagnosed with non metastatic breast cancer
* Candidate for mastectomy or breast-conserving surgery

Exclusion Criteria

* Patients with invasive tumors
* Patients receiving anti-cancer treatment
* Patients who have undergone surgery

Other protocol-defined exclusion criteria may apply.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Clinical response at 24 weeks

SECONDARY OUTCOMES:
Clinical response at 16 weeks
Clinical benefit at 16 weeks
Clinical benefit at 24 weeks
Rate of breast conserving surgery in both arms
Rate of complete pathological response
Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (10):
- Canada (10):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Granby, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Victoriaville, Quebec

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716